CLINICAL TRIAL: NCT00906295
Title: Establishment of Optimal Transfusion Threshold After Major Orthopedic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: TrygFonden, Denmark (Industry)
Responsible Party: MD Kamilla Nielsen, Rigshospitalet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-D-2009-024
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Last update posted 2011-06-06 (Estimated); Status verified 2011-06

CONDITIONS: Anemia; Arthroplasty; Replacement; Hip
Keywords: Hemoglobin; Ambulation
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Allowed drop in hemoglobin to 4.5-5.5 mmol/L (Active Comparator): Transfusion with red blood cells to level between 4.5-5.5 mmol/L
  Interventions: Other: Allowed drop in hemoglobin to 4.5-5.5 mmol/L
- Allowed drop in hemoglobin to 5.6-6.5 mmol/L (Experimental): Transfusion with red blood cells to level between 5.6-6.5 mmol/L
  Interventions: Other: Allowed drop in hemoglobin to level between 5.6-6.5 mmol/L

INTERVENTIONS:
Other: Allowed drop in hemoglobin to 4.5-5.5 mmol/L — Transfusion with red blood cells to hemoglobin between 4.5-5.5 mmol/L (Transfusion threshold of 4.5 mmol/L)
  Arms: Allowed drop in hemoglobin to 4.5-5.5 mmol/L
Other: Allowed drop in hemoglobin to level between 5.6-6.5 mmol/L — Transfusion with red blood cells to between hemoglobin 5.6-6.5 mmol/L (Transfusion threshold of 5.5 mmol/L)
  Arms: Allowed drop in hemoglobin to 5.6-6.5 mmol/L

SUMMARY:
The purpose of this study is to determine whether a higher threshold for transfusion with red blood cells improves the postoperative ambulation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Patients undergoing replacement of hip arthroplasty
* Be legally competent
* Read and understand Danish

Exclusion Criteria:

* Present malignant disease
* Known heart disease with functionality equivalent to NYHA II or CCS II or worse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go-test (TUG)in seconds. | 30 days
  Timed Up and Go-test is performed when the patient is able to undertake the test after surgery. This is judged by a physiotherapist. The test measures how long it takes the patient to rise, walk 3 meters, turn around, walk back and sit down again.

SECONDARY OUTCOMES:
The postoperative day patients can walk ten meters | 30 days
Length of stay at hospital | 30 days
The day the patient is able to perform Timed Up and Go-test | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Kamilla Nielsen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Bispebjerg Hospital, Copenhagen, Copenhagen NV
  - Copenhagen University Hospital, Rigshospitalet, Copenhagen, Østerbro

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836
- [Derived] Nielsen K, Johansson PI, Dahl B, Wagner M, Frausing B, Borglum J, Jensen K, Sturup J, Hvolris J, Rasmussen LS. Perioperative transfusion threshold and ambulation after hip revision surgery--a randomized trial. BMC Anesthesiol. 2014 Oct 10;14:89. doi: 10.1186/1471-2253-14-89. eCollection 2014. PMID 25337035
- See also: Official hospital homepage — http://www.rigshospitalet.dk